CLINICAL TRIAL: NCT04304846
Title: Attachment Representations of Children Born Prematurely in the Loire Infant Follow-up Team Cohort
Brief Title: AttachMent Preterm in the Loire Infant Follow-up Team
Acronym: AMPLIFy
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 49RC19_0132
Record Dates: First submitted 2020-03-10; First posted 2020-03-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Preterm Birth
Keywords: Prematurity; Attachment
MeSH Terms: conditions — Premature Birth | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AMPLIFy group: Mother, premature child and teacher will complete questionnaires and interviews on attachment, maternal stress and child behavior
  Interventions: Other: Questionnaires and interviews

INTERVENTIONS:
Other: Questionnaires and interviews — List of questionnaires: ASQ, PSI, PPQ, SDQ, GSA and AMMI score obtained from mother during two separated interviews for the mother and the child at 3 and 5 years old

SUMMARY:
The purpose of this study is to describe the attachment representations of children born prematurely at age 3 and 5 with regard to their neurocognitive and behavioral development.

DETAILED DESCRIPTION:
Whether they are born at term or prematurely, from birth, children seek contact with caregivers and establish privileged relationships with them. These attachment relationships are gradually established and, from the end of the first year, interindividual differences can be observed according to temperament, quality of interactions with adults and responses to children's needs for proximity and comfort.

Prematurity is a situation that can disrupt parent-child interactions. The physiological characteristics of the premature infant attenuate and distort his/her stress signals. Visual interactions are shorter, alertness is more labile and reactivity is less clear than that of babies born at term. In such situations of stress and trauma, maternal sensitivity and responsiveness can be affected. In addition, changes in the quality of mother-child interactions have been reported, with more controlling maternal behavior. This maternal trend has been associated with behavioral disorders in children, such as eating disorders or lack of interest in social communication. More frequent disruptions of maternal caregiving associated with relational withdrawal in the child have also been shown in the case of prematurity.

We hypothesize that the experience of establishing relationships with parents in a context of extreme prematurity can alter the development of secure attachment representations in the child and that maternal representations and their possible interactions with prematurity factors prevent or contribute to the development of insecure or disorganized attachment in the child. We also hypothesize that disorganized attachment representations are associated with somatic, environmental, affective, and neurodevelopmental complications (motor, cognitive and behavioral).

ELIGIBILITY:
Inclusion Criteria:

* Children born in the neonatal reanimation department of Angers and Nantes University Hospitals
* Extrem preterm infants (term of birth less than or equal to 28 weeks of amenorrhea)
* Children included in the regional monitoring network for vulnerable newborns (Réseau Grandir Ensemble en Pays de la Loire, RGE)
* Children with a follow-up consultation at age 3 scheduled as part of the classic RGE follow-up on the Angers and Nantes University Hospitals
* Informed consent dated and signed by the parents or the holder of the parental authority
* Affiliated to a Social Security scheme

Exclusion Criteria:

* Child with severe neurocognitive impairment or severe autism trait-type behavioral disorder in the 2-year RGE follow-up evaluation

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children born prematurely in the French region Pays de la Loire and included in the cohort 'Réseau Grandir Ensemble en Pays de la Loire'.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-01-07 (Actual); Primary Completion 2025-01-06 (Estimated); Study Completion 2027-01-06 (Estimated)

PRIMARY OUTCOMES:
Attachment Story Completion Task | Three and five years after preterm birth
  The evaluation of attachment representations will be realized at two stages of development, using attachment story stems to complete (Attachment Story Completion Task; Bretherton, Ridgeway & Cassidy, 1990), which is the gold standard tool for measuring this variable between the ages of 3 and 7. Four scores measuring security, deactivation, hyperactivation and disorganization are obtained with the coding system described by Miljkovitch (Miljkovitch et al. 2003). Score on each scale vary from -1 to +1.

SECONDARY OUTCOMES:
Attachment Multiple Model Interview (AMMI) | Three and five years after preterm birth
  The AMMI is a semi-structured interview, which assesses attachment representations regarding specific relationships including relationships with mother, father, and romantic partners (Miljkovitch, Moss, Bernier, Pascuzzo, & Sander, 2015). Scores vary from 0 to 8 for the security, deactivation, and hyperactivation scales and from 0 to 16 for the disorganization.
Parenting Stress Index (PSI) Scale | Three and five years after preterm birth
  The PSI is a 120-item self-report questionnaire assessing parenting stress in two main domains: The Parent Domain (51 items) measures stress related to parental functioning, the Child Domain (50 items) measures child qualities and characteristics that contribute to stress in the parent-child system. The PSI contains an additional Life Stress scale (19 items), which will not be used in the study. Scores vary from 50 to 250 in the Parent Domain and from 51 to 255 in the Child Domain. In both domains, higher scores indicate more stress.
Post-traumatic stress disorder Questionnaire (PPQ) | Three and five years after preterm birth
  A 14-item self-report questionnaire assessing the level of mothers' post-traumatic stress. A score between 0 and 56 is calculated.
Ages and Stages Questionnaires® (AQS) Questionnaires | Three and five years after preterm birth
  The ASQ-3 (and ASQ-5) assess 5 aspects of child development: communication, gross motor skills, fine motor skills, problem solving, and personal-social skills. Each aspect is evaluated through 6 questions. If the answer is yes, score = 10, sometimes = 5 and not yet = 0. The total scores obtained with the ASQ-3 and ASQ-5 range from 0 to 300.
Strengths and Difficulties Questionnaire (SDQ) | Three and five years after preterm birth
  The SDQ is a brief parent-report behavioral screening questionnaire for 3-16 year olds. It comprises 20 items relative to 5 categories: emotional problems, conduct problems, hyperactivity/inattention, peer relationship problems and prosocial behavior. The total score obtained with the SDQ is comprised between 0 and 50.
Global School Adaptation (GSA) Score | Five years after preterm birth
  The GSA score is an instrument designed for teachers to assess children's abilities and behavior in the classroom with 20 questions. Six questions investigate linguistic competence, five questions investigate non-verbal abilities, eight questions address children's behavior in the classroom and the final question invites the teacher to give his/her prognosis of the child's future adaptation to school life. Total scores vary from 20 to 60.

CONTACTS AND LOCATIONS:
Overall Officials: Elise Riquin, MD, Principal Investigator — University Hospital of Angers; Géraldine Gascoin, MD, Study Director — University Hospital of Angers
Locations (2):
- France (2):
  - University Hospital of Angers, Angers
  - University Hospital of Nantes, Nantes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Riquin E, Sandnes R, Bacro F, Vinay A, Miljkovitch R, Rouger V, Rakotonjanahary J, Gascoin G, Muller JB. A Prospective Observational Study to Assess Attachment Representations With Regard to Neurocognitive and Behavioral Outcomes in Children Born Very Prematurely in the Loire Infant Follow-Up Team (LIFT Cohort). Front Pediatr. 2022 Jul 13;10:896103. doi: 10.3389/fped.2022.896103. eCollection 2022. PMID 35903159